CLINICAL TRIAL: NCT03798665
Title: A Prospective, Multicenter, Non-interventional Registry Study Evaluating the Clinical Application of PEG-rhG-CSF During Chemotherapy in Patients With Malignant Solid Tumors in Sichuan
Brief Title: A Real World Study Evaluating the Clinical Application of PEG-rhG-CSF During Chemotherapy in Patients With Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Principal Investigator, DaiYuan Ma, Director of Cancer Center Affiliation: Afﬁliated Hospital of North Sichuan Medical College, Afﬁliated Hospital of North Sichuan Medical College
Other Study IDs: CB-RWS
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Neutropenia
MeSH Terms: conditions — Neutropenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pegfilgrastim（PEG-rhG-CSF） — From the first chemotherapy cycle using PEG-rhG-CSF (which can be any chemotherapy cycle of the patient), record the use of PEG-rhG-CSF in this cycle and each subsequent chemotherapy cycle, including dosage, administration time and dosing frequency

SUMMARY:
Prospective, multicenter, non-interventional registration studies were used in this project . Eight hundreds patients with solid tumors who met the inclusion criteria in six hospitals in Sichuan Province, Sichuan Province, were selected from the first chemotherapy cycle using PEG-rhG-CSF (can be any chemotherapy cycle of the patient), and each subsequent chemotherapy cycle was recorded. The use of PEG-rhG-CSF and related patient outcomes until the end of chemotherapy. Analyze the clinical practice of using PEG-rhG-CSF in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Diagnosed as a malignant solid tumor by histology and cytology, requiring chemotherapy patients;
3. The first use of PEG-rhG-CSF during the chemotherapy cycle (not limited to the first chemotherapy cycle, can be any chemotherapy cycle of the patient);
4. Subjects volunteered to participate in this clinical trial and signed informed consent.

Exclusion Criteria:

1. PEG-rhG-CSF was used in the current chemotherapy cycle;
2. Have received hematopoietic stem cell transplantation or bone marrow transplantation;
3. Other drug clinical trials are currently underway.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Age ≥ 18 years old;
  2. Diagnosed as a malignant solid tumor by histology and cytology, requiring chemotherapy patients;
  3. The first use of PEG-rhG-CSF during the chemotherapy cycle (not limited to the first chemotherapy cycle, can be any chemotherapy cycle of the patient);
  4. Subjects volunteered to participate in this clinical trial and signed informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-07-06 (Actual); Primary Completion 2019-07-06 (Estimated); Study Completion 2019-07-06 (Estimated)

PRIMARY OUTCOMES:
Dosage of PEG-rhG-CSF in chemotherapy | 1 YEAR
Administration time of PEG-rhG-CSF in chemotherapy | 1 YEAR
dosing frequency of PEG-rhG-CSF in chemotherapy | 1 YEAR

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan, China